CLINICAL TRIAL: NCT05850754
Title: American Veterans 4 Week Cannabidiol Intervention
Brief Title: 4 Week Veterans Cannabidiol Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Responsible Party: Principal Investigator, Laura Stewart, Professor, University of Northern Colorado
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2302048298
Record Dates: First submitted 2023-03-14; First posted 2023-05-09 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: cannabidiol; veterans; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to 1 of 2 groups and followed throughout a 4 week intervention period.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD Capsule (Experimental): Participants will take capsules containing 50 mg of CBD daily for 4 weeks.
  Interventions: Dietary Supplement: Vantage Hemp CBD
- Placebo Capsule (Placebo Comparator): Participants will take placebo capsules containing 0 mg of CBD daily for 4 weeks.
  Interventions: Dietary Supplement: Vantage Hemp Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Vantage Hemp CBD — Participants will consume 1 Vantage Hemp capsule, daily for 4 weeks.
  Arms: CBD Capsule
Dietary Supplement: Vantage Hemp Placebo Capsule — Vantage Hemp Placebo Capsule Intervention
  Arms: Placebo Capsule

SUMMARY:
Cannabidiol (CBD), a non-psychoactive hemp derivative, is an attractive therapeutic agent, and is most supported by the scientific community as an antiepileptic. Additionally, CBD is also associated with claims related to improvements in overall health, pain, anxiety, depression, and sleep; however, the scientific evidence is lacking. The overarching goal of this investigation is to determine the effects of a 4-week CBD intervention on measures of overall health, pain, anxiety, depression, and sleep in a population of US veterans. Primary aims will explore the effects of 4 weeks of CBD on pain, anxiety, and depression. Secondary aims will determine whether 4 weeks of CBD will affect general measures of overall health and sleep.

DETAILED DESCRIPTION:
In this double-blind investigation, participants will undergo 6 online assessments. Two assessments (assessments 1 and 2) will take place before the intervention period and assessments 3-6 will be conducted at the end of every week during the intervention period (assessment 3 at the end of week one, assessment 4 at the end of week 2, assessment 5 at the end of week 3 and assessment 6 at the end of week 4).

After participants (N=100) reach out to inquire about the study, they will be provided with an informed consent, and they will be asked to obtain physician approval to participate in the study. Once this approval is obtained, they will be randomized into either a cannabidiol ingesting group (CG, n=50, 50 mg of CBD per day)) or a placebo-controlled group (PC, n=50, 0 mg of CBD per day). Then, they will be sent a link to a survey which includes questions evaluating overall health, anxiety, depression, pain and sleep. The details of these surveys are outlined below. Once researchers receive a completed assessment 1, the participants will be mailed packages containing bottles of either CBD or a placebo capsules (32 capsules provided in each bottle). One week after assessment 1, participants will complete assessment 2 and will begin to take one capsule per day in the evening after their last meal. Participants will take the same online surveys in all assessments with the exception of the initial informed consent (in visit one only) as well as a few open-ended study experience questions in assessment 6. During the intervention period, all participants will complete capsule logs in which they confirm that they have consumed one of their assigned capsules each day. Subjects will take a picture and email the log back to researchers at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Biological Sex: Males or Females, Gender Binary or Non-Binary
* Veteran: US Veterans currently residing in the continental United States
* Informed Consent: The capability and willingness to give online informed consent, to understand the exclusion criteria, and to accept that the randomized group assignment is required.
* Secure Internet Access: Ability to use an online platform and agreement to take surveys and communicate with the research team while on a private (not public) device and using a private (not public) connection.

Exclusion Criteria:

* Pregnancy or Planned Pregnancy: Individuals who are pregnant or who are planning to become pregnant.
* Allergy to Capsule Ingredients: Individuals with a known allergy to porcine gelatin, glycerin, medium chain triglycerides (coconut derived), or CBD.
* Significant Mental Health Challenges: Presence of moderate to severe mental health challenges including paranoia, manic depression, bipolar disorder, severe depression or who are at risk for suicide.
* Significant Health Challenges: Presence of an uncontrolled chronic disease (heart disease, cancer, type 2 diabetes, etc) and/or individuals who are regularly taking anti-seizure drugs, blood thinners, antidepressants, anti-inflammatory drugs, muscle relaxants, sedatives, beta and calcium channel blocker and chemotherapy drugs, HIV antivirals. Individuals with seizure disorders.
* Illegal Substance Use: Individuals who are currently using illegal drugs.
* Cannabis or CBD Use: Individuals who have used a cannabis or CBD product(s) within the last 3 months.
* Residing in a State With CBD Restrictions: Residents of Idaho, Iowa, Missouri, South Dakota, Maine, and Nevada are not able to participate in this study.
* Travel Plans: Plans to travel outside of the continental United States during the 4 week study intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Veterans RAND 12 Item Health Survey single domains | Twice, separated by 1 week, prior to the start of the intervention and weekly during the 4 week intervention
  Veterans Health Survey RAND (VR-12). Two z scores are reported (Mental Component and Physical Component Scores)patient self-report, 12 questions, minimum value: 12 points, maximum value: 54 points, physical and mental health component summary score compared to a t-score with a mean value of 50 and standard deviation of 10
Change in General Anxiety Disorder Questionnaire Score | Twice, separated by 1 week, prior to the start of the intervention and weekly during the 4 week intervention
  General Anxiety Disorder Questionnaire 7.The GAD-7 scale score ranges from 0 to 21 points. A higher score suggests higher levels of anxiety.
Change in Beck Depression Inventory Score | Twice, separated by 1 week, prior to the start of the intervention and weekly during the 4 week intervention
  Beck Depression Inventory (BDI). Highest score is 63, Lowest score is 0.The higher the score, the more presence of depression.
Change in Defense and Veterans Pain Rating Scale Score | Twice, separated by 1 week, prior to the start of the intervention and weekly during the 4 week intervention
  Defense and Veterans Pain Rating Scale. Each item is scored 0 (no pain) - 10 (pain as bad as it can be). The higher the score indicates higher levels of pain.
Change in Pittsburg Sleep Quality Index Score | Twice, separated by 1 week, prior to the start of the intervention and weekly during the 4 week intervention
  Pittsburg Sleep Quality Index. Scores for each question range from 0-3. Higher scores indicating lower sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Stewart, PhD, Principal Investigator — University of Northern Colorado
Locations (1):
- University Of Northern Colorado, Greeley, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will become available when the study is published and will be available for 3 years.
Supporting Information: Study Protocol
Time Frame: Data will become available when the study is published and will be available for 3 years.
Access Criteria: Data (without subject ID numbers) will be shared upon email request laura.stewart@unco.edu.